CLINICAL TRIAL: NCT03011398
Title: Interventional Orthopedics Foundation Patient Registry Database-A Clinical Registry of Orthobiologics Procedures
Brief Title: A Clinical Registry of Orthobiologics Procedures
Status: Enrolling by invitation | Type: Observational
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RSI2015-REG01
Record Dates: First submitted 2016-12-29; First posted 2017-01-05 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Orthobiologic Procedures — To observe the improvement in subject-reported clinical outcomes for percutaneous orthopedic procedures used to treat musculoskeletal disorders.

SUMMARY:
The purpose of the Registry study is to observe the improvement in subject-reported clinical outcomes for percutaneous orthopedic procedures for treatment of musculoskeletal disorders.

DETAILED DESCRIPTION:
This Registry was designed to assure that the benefits and knowledge gained by studying clinical outcomes associated with the use of percutaneous orthopedic procedures outweigh the potential risks to the patients. The primary objective of this Registry is to observe the improvements in subject-reported clinical outcomes for these procedures used to treat musculoskeletal disorders. Secondary objectives include evaluating post-treatment complication, adverse events, re-injections, and surgical intervention. Patients receiving percutaneous orthopedic treatments are asked to enroll before receiving treatment and complete a set of baseline questionnaires regarding pain and functionality of the area of the body being treated (i.e. knee, shoulder, spine, etc). Follow-up outcomes are collected at 1 month, 3 months, 6 months, 12 months, 18 months, and annually 2-20 years post-injection. Subjects are withdrawn from the Registry prematurely if a surgical operation occurs.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must meet ALL of the following:

  1. Voluntary signature of the IRB approved Informed Consents,
  2. Treated with a Regenexx procedure
  3. Have a musculoskeletal condition appropriate for the procedure such as osteoarthritis or internal joint derangement; ligament or tendon injury; intervertebral disc degeneration; protrusion, extrusion, or annular tear; muscle tear

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with orthobiologics procedures
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2036-02 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Improvement | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean improvement score, where -100=100% worse from baseline and 100=100% better or improved from baseline

SECONDARY OUTCOMES:
Pain Scale | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean numeric pain score, where 0=no pain and 10=worst possible pain.
International Knee Documentation Committee form | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean IKDC score, where 0=lowest level of knee function and 100=highest level of knee function.
Lower Extremity Function Scale | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Means LEFS score, where 0=very low function of the lower extremity and 80=very high function of the lower extremity
Disabilities of the Arm, Shoulder and Hand form | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean DASH score, where 0=no disability of the upper extremity and 100=most severe disability of the upper extremity.
Oxford Hip Score | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean OHS score, where 42-48=excellent, 34-41=good, 27-33=fair, 0-26=poor for hip pain and function.
Functional Rating Index | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Mean FRI score, where 0=no disability in function of the neck and back and 100=severe disability.
Complications | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Description of any medical complication related to receiving a treatment procedure
Adverse Events | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Description of adverse events occurring after treatment procedure
Number of Re-injections to treated area | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  number of additional injections to treated area such as platelet rich plasma or stem cell treatment
Number of Surgical Interventions to treated area | 1 month, 3 months, 6 months, 12 months, 18 months and annually 2-20 years post treatment
  Number of surgical interventions to treated area after receiving treatment procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Regenerative Sciences, LLC and Centeno-Schultz Clinic
Locations (32):
- United States (30):
  - Catalyst Pain Solutions, Phoenix, Arizona
  - Healthlink Center, Beverly Hills, California
  - Healthlink Center, Oceanside, California
  - Healthlink Center, San Rafael, California
  - Southern California Orthopedic Institute, Thousand Oaks, California
  - Southern California Orthopedic Institute-Van Nuys, Van Nuys, California
  - Centeno-Schultz Clinic, Broomfield, Colorado
  - Regenexx, Broomfield, Colorado
  - New reGeneration Orthopedics, Sarasota, Florida
  - Chicago Arthritis, Chicago, Illinois
  - Orthopedic Stem Cell Resource, Des Plaines, Illinois
  - Harbor View Medical, Des Moines, Iowa
  - Bodyworks Musculoskeletal Medicine, Louisville, Kentucky
  - Total Care-LA, Lafayette, Louisiana
  - Stem Cell ARTS-MD, Chevy Chase, Maryland
  - RejuvMedical, Waite Park, Minnesota
  - New Jersey Sports Medicine, Cedar Knolls, New Jersey
  - Orthopedic Stem Cell Solutions, Oakhurst, New Jersey
  - Rehabilitation Center of New Jersey, Wayne, New Jersey
  - Rehabilitation Center of New York, New York, New York
  - Beacon Orthopaedics, Cincinnati, Ohio
  - ProMedica, Toledo, Ohio
  - RegenOrthoSport, Tulsa, Oklahoma
  - Columbia Pain Management, Hood River, Oregon
  - Rehabilitation and Pain Specialists, Pittsburgh, Pennsylvania
  - Center for Sports Medicine, Springfield, Pennsylvania
  - RegenOrthoSport, Dallas, Texas
  - Wasatch Pain Solutions, South Jordan, Utah
  - Vermont Regenerative Medicine, Winooski, Vermont
  - Stem Cell ARTS-VA, McLean, Virginia
- Nepean Specialist Sports Medicine, Kingswood, New South Wales, Australia
- RegenOrthoSport, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centeno CJ, Schultz JR, Cheever M, Robinson B, Freeman M, Marasco W. Safety and complications reporting on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2010 Mar;5(1):81-93. doi: 10.2174/157488810790442796. PMID 19951252
- [Background] Centeno CJ, Schultz JR, Cheever M, Freeman M, Faulkner S, Robinson B, Hanson R. Safety and complications reporting update on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2011 Dec;6(4):368-78. doi: 10.2174/157488811797904371. PMID 22023622
- [Background] Bain BJ. Morbidity associated with bone marrow aspiration and trephine biopsy - a review of UK data for 2004. Haematologica. 2006 Sep;91(9):1293-4. PMID 16956842
- [Background] Nejadnik H, Hui JH, Feng Choong EP, Tai BC, Lee EH. Autologous bone marrow-derived mesenchymal stem cells versus autologous chondrocyte implantation: an observational cohort study. Am J Sports Med. 2010 Jun;38(6):1110-6. doi: 10.1177/0363546509359067. Epub 2010 Apr 14. PMID 20392971
- [Background] Wakitani S, Okabe T, Horibe S, Mitsuoka T, Saito M, Koyama T, Nawata M, Tensho K, Kato H, Uematsu K, Kuroda R, Kurosaka M, Yoshiya S, Hattori K, Ohgushi H. Safety of autologous bone marrow-derived mesenchymal stem cell transplantation for cartilage repair in 41 patients with 45 joints followed for up to 11 years and 5 months. J Tissue Eng Regen Med. 2011 Feb;5(2):146-50. doi: 10.1002/term.299. PMID 20603892
- [Derived] Centeno CJ, Berger DR, Money BT, Dodson E, Urbanek CW, Steinmetz NJ. Percutaneous autologous bone marrow concentrate for knee osteoarthritis: patient-reported outcomes and progenitor cell content. Int Orthop. 2022 Oct;46(10):2219-2228. doi: 10.1007/s00264-022-05524-9. Epub 2022 Aug 6. PMID 35932306
- [Derived] Centeno CJ, Money BT, Dodson E, Stemper I, Steinmetz NJ. The rate of venous thromboembolism after knee bone marrow concentrate procedures: should we anticoagulate? Int Orthop. 2022 Oct;46(10):2213-2218. doi: 10.1007/s00264-022-05500-3. Epub 2022 Jul 18. PMID 35844014
- [Derived] Centeno C, Markle J, Dodson E, Stemper I, Williams C, Hyzy M, Ichim T, Freeman M. Symptomatic anterior cruciate ligament tears treated with percutaneous injection of autologous bone marrow concentrate and platelet products: a non-controlled registry study. J Transl Med. 2018 Sep 3;16(1):246. doi: 10.1186/s12967-018-1623-3. PMID 30176875
- [Derived] Centeno C, Markle J, Dodson E, Stemper I, Williams CJ, Hyzy M, Ichim T, Freeman M. Treatment of lumbar degenerative disc disease-associated radicular pain with culture-expanded autologous mesenchymal stem cells: a pilot study on safety and efficacy. J Transl Med. 2017 Sep 22;15(1):197. doi: 10.1186/s12967-017-1300-y. PMID 28938891